CLINICAL TRIAL: NCT03720860
Title: Prospective Studie of Inflammatory Markers in Urine, Plasma and Sputum Associated With Acute Kidney Injury
Brief Title: Inflammatory Mediators of Acute Kidney Injury in Intensive Care
Acronym: PronMed
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Robert Frithiof, MD, PhD, Uppsala University
Other Study IDs: 2017-043PronMed
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Surgery; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum Blood Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis: Patients admitted to the intensive care unit with sepsis
- Surgery: Patinets subjected to major surgery and then admitted to the intensive care unit
- Non-inflamed: Otherwise healthy patients admitted to the intensive care unit because of intoxication.

SUMMARY:
Acute kidney injury (AKI) affects more than 50% of patients admitted to the intensive care unit. The most common underlying cause is sepsis. Severe AKI in combination with sepsis is associated with high mortality. The mechanisms for sepsis-induced AKI are largely unknown. Our hypothesis is that the inflammatory response to an infection cause collateral damage to host tissue and contributes to the development of AKI. In this study we want to investigate the presence of novel inflammatory mediators in patients with sepsis, patients subjected to major surgery (sterile inflammation) and non-inflamed patients and correlate their levels with the risk for AKI.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the intensive/post operative care unit

* with septic shock or
* post major surgery or
* after intoxication with a chemical compund

Exclusion Criteria:

* Pregnancy or
* Breast feeding or
* Chronic kidney disease or
* intoxication with nephrotoxic compund or
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients subjected to major surgery or intensive care
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Histones | Within 1 month
  Correlation between levels of histones and degree of acute kidney injury

SECONDARY OUTCOMES:
Other inflammtory mediators | Within 1 month
  Correlation between levels of other inflammtory mediators and degree of acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska sjukhuset, Centraloperation, Uppsala, Uppsala County, Sweden